CLINICAL TRIAL: NCT02558634
Title: Thalamic Deep Brain Stimulation for Spasmodic Dysphonia: A Prospective, Randomized, Double-Blinded, Sham-Controlled Trial
Brief Title: Thalamic Deep Brain Stimulation for Spasmodic Dysphonia- DEBUSSY Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Neurosurgeon, Professor of Surgery (Neurosurgery), Director of Surgical Centre for Movement Disorders, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H15-02535
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Spasmodic Dysphonia; Laryngeal Dystonia; Deep Brain Stimulation
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS-on (Experimental): Ventral intermediate Nucleus (VIM) Thalamic DBS on
  DBS system includes:
  * Implantable Pulse Generator (IPG)
  * DBS Lead
  * DBS Lead Extension Kit
  Interventions: Device: VIM Thalamic Deep Brain Stimulation ON
- DBS-off (sham-stimulation) (Sham Comparator): Ventral intermediate Nucleus (VIM) Thalamic DBS off
  DBS system includes:
  * Implantable Pulse Generator (IPG)
  * DBS Lead
  * DBS Lead Extension Kit
  Interventions: Device: VIM Thalamic Deep Brain Stimulation OFF

INTERVENTIONS:
Device: VIM Thalamic Deep Brain Stimulation ON
  Arms: DBS-on
Device: VIM Thalamic Deep Brain Stimulation OFF
  Arms: DBS-off (sham-stimulation)

SUMMARY:
Laryngeal Dystonia (LD), also commonly referred to as spasmodic dysphonia, is a neurological voice disorder characterized by involuntary dystonic contractions of the laryngeal muscles. Current treatments such as botox and voice therapy only provide temporary relief and thus, the investigators are exploring new strategies to provide long-term, sustained improvement.

Deep Brain Stimulation (DBS) is a neurosurgical procedure that involves the implantation of electrodes to deliver electrical stimuli to specific brain regions. It is the standard surgical treatment for many other movement disorders such as Parkinson's disease, essential tremor, and primary dystonia. This trial has been designed to test the hypothesis that DBS can improve the vocal dysfunction of LD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed isolated laryngeal dystonia (adductor spasmodic dysphonia)
* Able to give informed consent
* Patients who fall into the age range of 18-75 years old
* Patients with inadequate medical and BTX management of spasmodic dysphonia

Exclusion Criteria:

* Dystonia present in other body parts (i.e- eyes, neck, limbs) in addition to larynx
* History of laryngeal denervation surgery for spasmodic dysphonia
* History of intracranial pathology (such as multiple sclerosis, tumors, or aneurysms) that may account for dystonia or essential tremor.
* History or evidence of ongoing psychiatric or neurodegenerative disorders (such as Parkinson's disease, Alzheimer's disease).
* Incompetent adults or those unable to communicate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Honey, MD, DPhil, Principal Investigator — UBC
Locations (1):
- The Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Ludlow CL, Adler CH, Berke GS, Bielamowicz SA, Blitzer A, Bressman SB, Hallett M, Jinnah HA, Juergens U, Martin SB, Perlmutter JS, Sapienza C, Singleton A, Tanner CM, Woodson GE. Research priorities in spasmodic dysphonia. Otolaryngol Head Neck Surg. 2008 Oct;139(4):495-505. doi: 10.1016/j.otohns.2008.05.624. PMID 18922334
- [Background] Simonyan K, Tovar-Moll F, Ostuni J, Hallett M, Kalasinsky VF, Lewin-Smith MR, Rushing EJ, Vortmeyer AO, Ludlow CL. Focal white matter changes in spasmodic dysphonia: a combined diffusion tensor imaging and neuropathological study. Brain. 2008 Feb;131(Pt 2):447-59. doi: 10.1093/brain/awm303. Epub 2007 Dec 14. PMID 18083751
- [Derived] Hart MG, Polyhronopoulos N, Sandhu MK, Honey CR. Deep Brain Stimulation Improves Symptoms of Spasmodic Dysphonia Through Targeting of Thalamic Sensorimotor Connectivity. Neurosurgery. 2024 Jan 22;94(6):1291-300. doi: 10.1227/neu.0000000000002836. Online ahead of print. PMID 38251897
- [Derived] Honey CR, Kruger MT, Almeida T, Rammage LA, Tamber MS, Morrison MD, Poologaindran A, Hu A. Thalamic Deep Brain Stimulation for Spasmodic Dysphonia: A Phase I Prospective Randomized Double-Blind Crossover Trial. Neurosurgery. 2021 Jun 15;89(1):45-52. doi: 10.1093/neuros/nyab095. PMID 33862624
- [Derived] Poologaindran A, Ivanishvili Z, Morrison MD, Rammage LA, Sandhu MK, Polyhronopoulos NE, Honey CR. The effect of unilateral thalamic deep brain stimulation on the vocal dysfunction in a patient with spasmodic dysphonia: interrogating cerebellar and pallidal neural circuits. J Neurosurg. 2018 Feb;128(2):575-582. doi: 10.3171/2016.10.JNS161025. Epub 2017 Mar 17. PMID 28304188

RESULTS

PARTICIPANT FLOW:
Groups:
- DBS-on First, Then DBS-off (Sham-stimulation): Ventral intermediate Nucleus (VIM) Thalamic DBS on for the first 3 months, then Thalamic DBS off for the next 3 months
  DBS system includes:
  * Implantable Pulse Generator (IPG)
  * DBS Lead
  * DBS Lead Extension Kit
  VIM Thalamic DBS ON for first 3 months, then Thalamic DBS OFF for following 3 months
- DBS-off First (Sham-stimulation), Then DBS-on: Ventral intermediate Nucleus (VIM) Thalamic DBS off (Sham-stimulation) for the first 3 months, then Thalamic DBS on for the following 3 months
  DBS system includes:
  * Implantable Pulse Generator (IPG)
  * DBS Lead
  * DBS Lead Extension Kit
  VIM Thalamic Deep Brain Stimulation OFF for first 3 months, followed by VIM Thalamic Deep Brain Stimulation ON for the following 3 months
Period: Blinded: First Intervention (3 Months)
Arm/Group | DBS-on First, Then DBS-off (Sham-stimulation) | DBS-off First (Sham-stimulation), Then DBS-on
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0
Period: Blinded: Second Intervention (3 Months)
Arm/Group | DBS-on First, Then DBS-off (Sham-stimulation) | DBS-off First (Sham-stimulation), Then DBS-on
Started | 4 | 2
Completed | 3 (Assessed after 2 weeks - 1 participant requested to have their DBS 'on') | 2
Not Completed | 1 | 0
Period: Unblinded: DBS on (6 Months)
Arm/Group | DBS-on First, Then DBS-off (Sham-stimulation) | DBS-off First (Sham-stimulation), Then DBS-on
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 1. Patients who are currently receiving BTX injections for their voice disorder
  2. Who experience fluctuations in their symptom control as a result of their BTX therapy
  3. Patients who fall into the age range of 18-75 years old
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.17 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6
Patients who are currently receiving BTX injections for their voice disorder [Count of Participants; unit: Participants] | 6
Patients who experience fluctuations in their symptom control as a result of their BTX therapy [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Unified Spasmodic Dysphonia Rating Scale (USDRS)
Description: Assessments of spasmodic dysphonia using a standardized spasmodic dysphonia rating scale were done pre-operatively, blinded DBS ON, blinded DBS OFF, and open DBS ON. Voice recording taken of each patient reading standardized sentences were blinded and evaluated by two speech language pathologists. The scale ranges from 0-7, with lower scores being better and higher scores being worse.
Time Frame: After the first 6 months, the participants completed the USDRS twice (once per crossover).
Population: One patient requested to have their DBS on after 2 weeks of being in the blinded-DBS OFF after the first crossover.
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Blinded-DBS ON: All participants who at some point in the study were in the 3-month blinded DBS ON intervention.
- Blinded-DBS OFF: All participants who at some point in the study were in the 3-month blinded DBS OFF intervention.
Arm/Group | Blinded-DBS ON | Blinded-DBS OFF
Number analyzed (Participants) | 6 | 5
units on a scale | 2.5 (1.4) | 3.75 (1.0)
Statistical Analysis 1: Comparison: Blinded-DBS ON; Test type: Superiority; p = 0.025, Wilcoxon (Mann-Whitney) — The level of significance was set at p=0.025 to allow a Bonferroni correction for these two tests (i.e. p=0.050 divided by two); Median Difference (Final Values) = 1.25, 95% CI 2-sided [0.75 to 1.75]

2. Primary Outcome: Voice-Related Quality of Life
Description: Double-blinded assessments of voice-related quality of life with DBS ON/OFF were conducted using the V-RQoL for Spasmodic Dysphonia. The V-RQoL is a questionnaire that measures a patient's voice related quality of life. The scale ranges from 0-50, with higher scores representing a lower quality of life with respect to voice.
Time Frame: After the first 6 months, the participants completed the V-RQoL twice (once per crossover).
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Blinded-DBS ON | Blinded-DBS OFF
Number analyzed (Participants) | 6 | 5
units on a scale | 74.7 (18.3) | 19 (18.2)

3. Secondary Outcome: Beck's Depression Inventory Scale
Description: Beck's Depression Inventory Scale (BDI-II) was used in this study to evaluate the mood of the patients both pre-operatively and at the end of the one-year study.
  All 6 patients completed the BDI-II, which is a scale that identifies symptoms and attitudes associated with depression, and evaluates the presence and severity of depression. The BDI-II ranges from 0-63. Scores ranging from 0-10 are considered to be absent or minimal depression, 10-18 indicate mild to moderate depression, 19-29 indicate moderate depression, and 30-63 indicate severe depression.
Time Frame: All participants completed the BDI-II once pre-operatively and once 1 year post-operatively (after the 6-month open unblinded phase).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-DBS ON: All participants in the study were assessed using the BDI-II pre-operatively and then again at the end of the 6-month open DBS ON phase (1 year post-op).
Arm/Group | Open-DBS ON
Number analyzed (Participants) | 6
units on a scale
  Pre-Operative BDI-II | 13.33 (7.20)
  One Year Follow-Up BDI-II | 6.50 (6.47)

4. Secondary Outcome: Montreal Cognitive Assessment Scale (MoCA)
Description: The MoCA was used to analyze the cognitive ability of the patients. It was first evaluated pre-operatively and again evaluated at the end of the one-year study. The MoCA scale ranges from 0-30 with higher scores indicating less cognitive impairment. Scores ranging from 18-25 indicate mild cognitive impairment, 10-17 indicate moderate cognitive impairment, and scores less than 10 indicate severe cognitive impairment.
Time Frame: All participants completed the MoCA once pre-operatively and once 1 year post-operatively (after the 6-month open unblinded phase).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-DBS ON: All participants in the study were assessed using the MoCA pre-operatively and then again at the end of the 6-month open DBS ON phase (1 year post-op).
Arm/Group | Open-DBS ON
Number analyzed (Participants) | 6
units on a scale
  Pre-Operative MoCA | 24.17 (3.08)
  One Year Follow-Up MoCA | 26.67 (3.09)

5. Secondary Outcome: Voice-Handicap Index
Description: The Voice-Handicap Index (VHI) is a questionnaire that measures the patients' perceived degree of handicap related to their voice. The VHI ranges from a scale of 0-100, with higher scores reflecting higher perceived degree of voice handicap and lower scores reflecting lower perceived degree of voice handicap.
Time Frame: All participants completed the VHI once pre-operatively and once 1 year post-operatively (after the 6-month open unblinded phase).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-DBS ON: All participants in the study were assessed using the VHI pre-operatively and then again at the end of the 6-month open DBS ON phase (1 year post-op).
Arm/Group | Open-DBS ON
Number analyzed (Participants) | 6
units on a scale
  Pre-Operative VHI | 84.83 (15.52)
  1 Year Post-Operative VHI | 38.17 (13.15)

ADVERSE EVENTS:
Time Frame: The study took place from January 1, 2017 - May 30, 2018. The study duration was approximately 1.5 years.
Description: This cohort continues to be followed and any future adverse events will be reported.
Groups:
- Blinded DBS-ON; Open DBS-ON: When DBS was turned on, none of the patients had any adverse clinical events during the trial. There were no asymptomatic hemorrhages detected on the post-operative CT scans. At the conclusion of the trial (1-year post-operative), there had been no infections, erosions, or technical malfunctions. The cohort continues to be followed and future adverse event will be reported.
- Blinded DBS-OFF: When DBS was turned off, none of the patients had any adverse clinical events during the trial. There were no asymptomatic hemorrhages detected on the post-operative CT scans. At the conclusion of the trial (1-year post-operative), there had been no infections, erosions, or technical malfunctions. The cohort continues to be followed and future adverse event will be reported.
Arm/Group | Blinded DBS-ON | Blinded DBS-OFF | Open DBS-ON
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT02558634/Prot_SAP_000.pdf